CLINICAL TRIAL: NCT04274179
Title: A Prospective, Case-control Evaluation of Ketogenic Dietary Therapy for New-onset Childhood Absence Epilepsy
Brief Title: Ketogenic Diet for New-Onset Absence Epilepsy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00241856
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Absence Epilepsy; Ketogenic Dieting; Epilepsy, Absence
Keywords: ketogenic; diet; absence
MeSH Terms: conditions — Epilepsy, Absence | interventions — Ethosuximide; Valproic Acid; Lamotrigine

STUDY DESIGN:
Intervention Model Description: Two arms (diet and drugs) with ability to cross-over at 1 or 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Diet therapy (Experimental): Modified Atkins Diet - high fat, low carbohydrate, outpatient initiated approach. Parents will check urine ketones twice weekly and follow by email, phone and clinic. Labs at baseline and 3 months. Dietitian support.
  Interventions: Other: Modified Atkins Diet
- Drug therapy (Active Comparator): Families will have the usual care for absence epilepsy at the discretion of the family's neurologist and the family choice. Typically ethosuximide bis in die (BID), however, if convulsions have occurred or other factors are involved, the child may be started on valproate or lamotrigine. The child will continue medications with dose adjustment and antiseizure drug levels checked as usual. **OF NOTE, THIS ARM IS COMPLETED
  Interventions: Drug: Absence epilepsy medications

INTERVENTIONS:
Other: Modified Atkins Diet — Low carb (20g/day), high fat, moderate protein diet. Started as an outpatient in clinic.
  Arms: Diet therapy
Drug: Absence epilepsy medications — At neurologist's discretion. *OF NOTE< THIS ARM IS COMPLETED
  Other Names: Ethosuximide, valproate or lamotrigine
  Arms: Drug therapy

SUMMARY:
The ketogenic diet is a medical therapy for epilepsy that is used nearly predominantly for refractory epilepsy (after 2-3 drugs have been tried and failed). However, there is both published evidence for first-line use (infantile spasms, Glut1 deficiency syndrome) and also anecdotal experience (families choosing to change the child's (or the family' own) diet rather than use anticonvulsant medications). Childhood absence epilepsy (refractory) has been published as being responsive to ketogenic diet therapy by the investigators' group previously. This is a small, prospective, 3 month trial to assess if using a modified Atkins diet is a feasible and effective option for new-onset childhood absence epilepsy. The investigators will compare to a group of children in which the parents have declined and chose to start anticonvulsant medications.

DETAILED DESCRIPTION:
The ketogenic diet has been in continuous use since 1921 for children and adult with medically-refractory epilepsy. One of the major unanswered questions is whether it would be as effective for children with new-onset epilepsy. Although logically, this would be the case, it remains to be shown in clinical trials. Additionally, it is much easier to take a medication than to change dietary habits and there is doubt whether families would truly wish to try dietary therapy first (or stay on dietary therapy if not effective for a 6 month trial period).

There is limited published evidence supporting the use of the ketogenic diet as a first-line therapy for infantile spasms, myoclonic astatic epilepsy, and in some situations where a family member had success and the family wishes to start it first. However, these are relatively rare conditions. The emergence of the modified Atkins diet as an outpatient, quickly-initiated, non-fasting approach since 2003 has changed the concept of dietary therapy towards a much less restrictive, potentially emergent therapy. In this way, using dietary therapy could potentially be started before medications for a willing family.

The use of dietary therapy (including the modified Atkins diet) for childhood absence epilepsy goes back decades, but was recently profiled in a review article from the investigators' group. In this publication, 17 studies were identified, and 69% of 133 children with refractory childhood absence epilepsy had a >50% seizure reduction and 34% were seizure-free. At the investigators' center, 21 children as of 2011 had been treated with dietary therapy with 19% seizure-freedom. The question of whether results would be similar (or better) for children with new-onset absence epilepsy was unanswered.

The standard treatments for childhood absence epilepsy (ethosuximide, valproate, lamotrigine) are effective in ~50% of children by 16-20 weeks. However, side effects exist and include stomach upset, inattention, mood disturbance, rash, liver function test abnormalities, and fatigue. Families at times do ask about avoiding treatment completely, especially as this epilepsy usually resolves in puberty and convulsions only occur in 20% (most children have brief staring spells only). In addition, families do also ask about "nonpharmacologic" treatment, but to date the investigators have not recommended it due to lack of data.

This study will have 20 children in each arm (diet and drug) with ability to crossover. Parents with a child with new-onset absence epilepsy will choose between the two therapies. Visits will be at baseline, 1 month and 3 months. EEG, labs and clinic visits will be paid by the parent's insurance (not free).

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3-12 years at seizure onset with classic childhood absence epilepsy clinically.
* Normal intellect or mild disability
* EEG with confirmed 3/second spike-wave discharges, usually with hyperventilation
* Daily reported absence seizures.
* Generalized convulsions allowed

Exclusion Criteria:

* Previous treatment with any anticonvulsant drug
* Previous use of a ketogenic dietary therapy for epilepsy or any other condition
* Glut1 deficiency syndrome
* Metabolic disorder known that would preclude dietary therapy
* Dietary restrictions for which a high fat, low carbohydrate diet would be precluded.
* Prior history of epilepsy (febrile seizures allowed)
* Unwilling to consent to study procedures or return for visits

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in seizure frequency | At 1 and 3 months post treatment
  Parental report of seizure frequency.

SECONDARY OUTCOMES:
Tolerability of diet therapy as assessed by restrictiveness of the diet therapy | At 3 months
  Diet therapy restrictiveness will be assessed with an open ended questionnaire that asks "how hard has it been for the child?". Completely subjective with no scale or scoring.
Tolerability of diet therapy as assessed by restrictiveness of the diet therapy | At 6 months
  Diet therapy restrictiveness will be assessed with an open ended questionnaire that asks "how hard has it been for the child?". Completely subjective with no scale or scoring.
Duration of diet therapy | Up to 3 months post treatment
  Duration of diet therapy in months.
Tolerability of diet therapy as assessed by change in urinary ketones | At 1 and 3 months post treatment
  Urinary ketones in mg/dl will be measured (80-160mg/dl is considered large ketosis).
EEG changes (normalization of the baseline spike-wave bursts) | Baseline and at 3 months post treatment
  30 minute routine EEG including hyperventilation to induce seizures, compare 3 months to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eric H Kossoff, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Groomes LB, Pyzik PL, Turner Z, Dorward JL, Goode VH, Kossoff EH. Do patients with absence epilepsy respond to ketogenic diets? J Child Neurol. 2011 Feb;26(2):160-5. doi: 10.1177/0883073810376443. Epub 2010 Jul 20. PMID 20647578
- [Background] Kossoff EH, Hedderick EF, Turner Z, Freeman JM. A case-control evaluation of the ketogenic diet versus ACTH for new-onset infantile spasms. Epilepsia. 2008 Sep;49(9):1504-9. doi: 10.1111/j.1528-1167.2008.01606.x. Epub 2008 Apr 10. PMID 18410363